CLINICAL TRIAL: NCT05660343
Title: Evaluation of the Efficacy of Ozonated Olive Oil and Low-Level Laser Therapy in the Treatment of Pain in Individuals With Temporomandibular Disorder
Brief Title: Ozonated Olive Oil and Low-Level Laser Therapy in TMD Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, levent Cigerim, Head of oral and maxillofacial department, Yuzuncu Yil University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17.06.2020/18
Record Dates: First submitted 2022-12-12; First posted 2022-12-21 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: TMD

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: In order to apply the principle of double-blind, we ensure that neither the laser therapist nor the patient knew whether the treatment was active or not, classical music was played in the background to mask the laser sound and the laser's programs were arranged by an assistant so that the treatment did not begin until a permission was taken from the assistant; in addition, labels on Oil bottles were removed by an assistant to ensure that no one knew the type of the Oil or its ingredients. For safety reasons, both the patient and the laser therapist wore protective goggles during the laser treatment. All patients were treated with ozonated olive oil and LLL by the same therapist.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ozonated olive oil (Experimental): (0.03PPM ozone + 6-6.5 PH olive oil, viscosity at 25°C 55mPas, relative density gr/ml (20°C) 0.98 pycnometer, Ozonated olive oil, 100 ml bottle, Olive Farm, GÜLLERDAĞI TURİZM TARIM İNŞ), Ozonated Olive Oil is used 3 times a day, every day for four weeks. Patients were instructed to spray three times on each side. To ensure commitment, Oil canisters were marked in the middle, which the patient was required to use until the label in the first two weeks, and the remaining amount in the second two weeks.
  Interventions: Drug: Ozonized Olive Oil Solutions
- Ozonated olive oil with low level laser therapy (Experimental): (810 nm diode laser, 3.4 j/cm2 energy density, 0.5w power, CHEESE DEN7A/DEN4A 810, 2 min for each side) was applied non-contact at a distance of 1 cm, the most painful points in the muscles diagnosed during the first examination were irradiated with circular movements and patients were called for 3 sessions per week over four weeks.
  Interventions: Drug: Ozonized Olive Oil Solutions; Device: Low Level Laser LLL Therapy

INTERVENTIONS:
Drug: Ozonized Olive Oil Solutions — (0.03PPM ozone + 6-6.5 PH olive oil, viscosity at 25°C 55mPas, relative density gr/ml (20°C) 0.98 pycnometer, 100 ml bottle.
Device: Low Level Laser LLL Therapy — (0.03PPM ozone + 6-6.5 PH olive oil, viscosity at 25°C 55mPas, relative density gr/ml (20°C) 0.98 pycnometer, Ozonated olive oil, 100 ml bottle, and 810 nm diode laser, 3.4 j/cm2 energy density, 0.5w power, CHEESE DEN7A/DEN4A 810, 2 min for each side
  Arms: Ozonated olive oil with low level laser therapy

SUMMARY:
The aim of the present study was to determine the efficacy of ozonated olive oil and low-level laser therapy (LLLT) in treating pain in individuals with TMD. In this prospective, randomized, split-mouth, double-blind study, two different treatment methods were applied to the patients.

DETAILED DESCRIPTION:
two different treatment methods were applied to the patients. Group 1 (study group, one side of the same patient): topical ozonated olive oil + LLLT; Group 2 (the other side of the same patient): Olive oil with topical ozone + LLLT (not activated). The ozonated olive oil was applied topically three times a day for four weeks, the LLLT was applied noncontact at a distance of 1 cm, and patients attended three sessions per week for four weeks. Before starting treatment, and after 6 sessions of laser therapy, the patients were evaluated. (2 weeks), after 12 laser sessions (1 month), and 3 months after the first session.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals aged 18 and over,
2. Individuals should be literate so that they can evaluate the consent form themselves,
3. Individuals with no restrictions to the use of any medication to be prescribed during the study,
4. Individuals who have not been treated for temporomandibular joint disease in the past 3 months,
5. Individuals who have not used any medication for the past two weeks,
6. Individuals who will participate in the study must be residing in the province of Van so that their regular records can be obtained,
7. Individuals without systemic disease,
8. Individuals with chronic pain, (pain that has been ongoing and lasted longer than six months),
9. Individuals with bilateral pain complaints,
10. Individuals without missing teeth,
11. Individuals without open bite and/or crossbite,

Exclusion Criteria:

1. Individuals with internal disorders and/or inflammatory joint disorders and/or joint's sound, 25
2. Individuals who have undergone interventional or surgical procedures on the Temporomandibular joint,
3. Individuals with temporomandibular joint pathology,
4. Individuals with the possibility of either being pregnant, are pregnant or lactating,
5. Individuals who will not attend postoperative check-ups,
6. Individuals using drugs other than those recommended,
7. Individuals who are allergic to any of the drugs and materials to be used throughout the study,
8. Individuals with contraindications to Ozone or Laser therapy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2020-06-17 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Pain Evaluation | Pre-treatment
  Patients will be requested to mark their pain intensity on a pain assessment form using a visual analog scale (VAS) ranging between 0 (no pain) to 10 (most severe pain).
Pain Evaluation | Post-treatment (after 2 weeks )
  Patients will be requested to mark their pain intensity on a pain assessment form using a visual analog scale (VAS) ranging between 0 (no pain) to 10 (most severe pain).
Pain Evaluation | Post-treatment (after 1 month)
  Patients will be requested to mark their pain intensity on a pain assessment form using a visual analog scale (VAS) ranging between 0 (no pain) to 10 (most severe pain).
Pain Evaluation | Post-treatment (after 3 months)
  Patients will be requested to mark their pain intensity on a pain assessment form using a visual analog scale (VAS) ranging between 0 (no pain) to 10 (most severe pain).

CONTACTS AND LOCATIONS:
Locations (1):
- Van Yüzüncü Yıl University, Van, Turkey (Türkiye)